CLINICAL TRIAL: NCT04112888
Title: Efficacy of Infiltrations With Collagen in Pelvic Pain Caused by Episiotomy and Cesarean Scars. Pilot Study
Brief Title: Infiltrations With Collagen in Episiotomy and Cesarean Scars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Althaia Xarxa Assistencial Universitària de Manresa (Other)
Responsible Party: Principal Investigator, Georgia Romero, Principal Investigator, Althaia Xarxa Assistencial Universitària de Manresa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEI 17/73
Record Dates: First submitted 2019-01-02; First posted 2019-10-02 (Actual); Last update posted 2019-10-02 (Actual); Status verified 2019-10

CONDITIONS: Pelvic Pain
Keywords: Episiotomy; Pain; Colagen
MeSH Terms: conditions — Pelvic Pain; Pain | interventions — Collagen

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Collagen group (Experimental): Patients will receive 3 to 5 infiltrations of collagen on the scar once a week.
  Patients will receive the conventional treatment of 8 rehabilitation sessions with massage therapy techniques, muscle stretches and fascial work. The rehabilitation sessions will always be carried out by the same physiotherapist specialized in pelvic floor. Two rehabilitation sessions per week during four weeks. The rehabilitation sessions will last 45 minutes.
  Interventions: Combination Product: Collagen; Procedure: Rehabilitation sessions
- Control group (Active Comparator): Patients will receive the conventional treatment of 8 rehabilitation sessions with massage therapy techniques, muscle stretches and fascial work. The rehabilitation sessions will always be carried out by the same physiotherapist specialized in pelvic floor. Two rehabilitation sessions per week during four weeks. The rehabilitation sessions will last 45 minutes.
  Interventions: Procedure: Rehabilitation sessions

INTERVENTIONS:
Combination Product: Collagen — Patients will receive 3 to 5 collagen infiltrations in the scar once per week. Patients with episiotomy will receive 3 collagen infiltrations while patients who underwent a cesarean section will receive 5 collagen infiltrations. The infiltration will be done by tunneling technique, that is, it will be applied along the scar, placing the needle almost tangential to the entire length of the area, then it will be injected and at the same time the needle will be removed. Infiltrations will be carried out intradermally, previously performing asepsis in the area to be infiltrated. 2 ml syringes will be used to infiltrate the episiotomy scars (we will use 1 vial of 2 ml ) and 5 ml for cesarean scars (2 vials of 2 ml ) and sterile needles of 30G, 13mm.
  Arms: Collagen group
Procedure: Rehabilitation sessions — Patients will receive the conventional treatment of 8 rehabilitation sessions with massage therapy techniques, muscle stretches and fascial work. The rehabilitation sessions will always be carried out by the same physiotherapist specialized in pelvic floor. There will be two sessions per week for four weeks. The sessions will last 45 minutes.

SUMMARY:
One of the causes of pelvic pain is secondary to scarring due to episiotomy or cesarean after delivery.The pain of episiotomies or cesarean scars can be generalized at the level of the perineum, or more specifically at the level of the scar. For all these reasons, the presence of painful scars after a delivery, either by a cesarean or an episiotomy produces a perception of pelvic pain and change is your body schema and a series of negative connotations such as secondary dyspareunia, affective alterations, etc.

To this, the investigators must add the important role that the psychological and social aspects can play in the development and perpetuation of a pain of these characteristics.

The perception of pain is subjective and its intensity will be perceived based on many variables in each individual. The psycho-corporal representation of the episiotomy and/or cesarean section and its consequences will depend on each woman. In addition to the physical aspect, the scar of the episiotomy is the testimony of the birth and its complications. It causes a change in the representation of the body and the sex of the patient.

The objective of this study is to evaluate the efficacy of collagen infiltrations in pelvic pain and the appearance of painful scars of episiotomies and/or cesareans compared to conventional treatment with rehabilitation.

DETAILED DESCRIPTION:
Randomized clinical trial to evaluate the efficacy of collagen infiltrations in pelvic pain caused by cesarean scars and/or episiotomies.

Those patients who are referred to the Rehabilitation consultation for pelvic pain secondary to pain in the cesarean/episiotomy scar who meet the inclusion criteria and who agree to participate and sign the informed consent will be included.

In the baseline assessment, the patient's clinical information will be collected: age, obstetric history, pathological history, active treatments and if they breastfeed. The following questionnaires will be passed: the Visual Analogue Scale (VAS) and the Short Form McGill Pain Questionnaire (SF-MPQ) to evaluate the pain caused by the scar, the Vancouver Scale of Healing (VSS) and the Patient Component (PSAS) of the Patient and Observer Objective Assessment Scale (POSAS) for the evaluation of the scar and initial photograph of the scar. A physical examination of the pelvic floor will be performed and the areas to be infiltrated will be detected.

Patients will be randomly assigned to a Control group, will perform the conventional treatment, and an Experimental Group, who will perform the conventional treatment and will also have 3-5 infiltrations with collagen.

At 6 and 16 weeks to finalize the treatment, a blinded assessor will perform the final assessment by passing the questionnaires used in the baseline assessment. The subjective satisfaction of the clinician and the patient will also be assessed using the questionnaires Clinical Global Improvement Impression Scale (GGI-I) and the Patient Global Improvement Impression Scale (PGI-I).

ELIGIBILITY:
Inclusion Criteria:

1. Patients between 18-45 years old.
2. Between 2 and 36 months post-partum
3. Accept participate in the study and sign the informed consent.

Exclusion Criteria:

1. Mental or cognitive disorder that prevents comprehension.
2. Being pregnant.
3. Pacemaker carriers.
4. On treatment with oral anticoagulants.
5. Local infections at the point of infiltration.
6. Total or partial denervation of the pelvic floor.
7. Neurological diseases: AVC, LM, MS.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2018-04-01 (Actual)

PRIMARY OUTCOMES:
Pain caused by the scar (VAS) | 6 weeks after the end of treatment
  Pain caused by the scar according to the Visual Analogue Scale (VAS). Range 0 to 10. Higher values represent worse pain.
Pain caused by the scar (MPQ) | 6 weeks after the end of treatment
  Pain caused by the scar according to the Short Form McGill Pain (Questionnaire (MPQ). Range 0 to 78. Three dimensions: Sensory (12 ítems), Affective (3 ítems), Evaluative (1 ítem). Higher score higher level of pain.

SECONDARY OUTCOMES:
Aspect of the scar (VSS) | 6 weeks after the end of treatment
  Aspect of the scar according to the Vancouver Scar Scale (VSS). Range 0 to 10. 0 (representing normal skin) and 10 (representing worst scar imaginable).
Aspect of the scar (PSAS) | 6 weeks after the end of treatment
  Aspect of the scar according to according to the patient component (PSAS) of the Scale of objective assessment Patient and Observer (Patient and Observer Scar Assesment Scale POSAS). The PSAS consist of six parameters: scar-related pain, itchness, color, stiffeness, thickness, and irregularity. Each parameter used a 10-point scoring system, with 1 representing normal skin and 10 representing the worst scar imaginable.
Subjective satisfaction of the clinician (PGI-I) | 6 weeks after the end of treatment
  Subjective satisfaction of the clinician according to Patient Global Impression of Im,provement (PGI-I). Single question asking the patient to rate their satisfaction now, as compared with how it was prior to before beginning treatment on a scale from 1-Very much better to 7 -Very much worse.
Subjective satisfaction of the clinician (CGI-I) | 6 weeks after the end of treatment
  Subjective satisfaction of the clinician according to Clinician Global Impression of Improvement (CGI-I). Single question asking the clinician to rate their satisfaction now, as compared with how it was prior to before beginning treatment on a scale from 1- Much better to 5-Much worse.

CONTACTS AND LOCATIONS:
Overall Officials: Georgia Romero-Culleres, MD, PhD, Principal Investigator — Althaia Xarxa Assistencial Universitària de Manresa
Locations (1):
- Althaia Xarxa Assistencial Universitària de Manresa, Manresa, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided